CLINICAL TRIAL: NCT01831791
Title: Study ARI114264: A Long-Term Study of the Safety and Efficacy of Dutasteride in the Treatment of Male Subjects With Androgenetic Alopecia
Brief Title: A Long-term Study to Determine Safety and Efficacy of Dutasteride in Male Subjects With Androgenetic Alopecia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114264
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Alopecia
Keywords: male pattern hair loss; hair growth; hair restoration; Dutasteride; Androgenetic alopecia; safety; efficacy
MeSH Terms: conditions — Alopecia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dutasteride Arm (Experimental): Subjects will receive 1 capsule of Dutasteride 0.5 mg orally once daily for 52 weeks (12 months).
  Interventions: Drug: Dutasteride 0.5 mg

INTERVENTIONS:
Drug: Dutasteride 0.5 mg — Dutasteride will be supplied as soft gelatin capsules, containing 0.5 mg of Dutasteride and it will be packaged in high-density polyethylene (HDPE) bottles with plastic child-resistant closures.

SUMMARY:
This is a multicentre, open-label study to assess the safety, tolerability, and efficacy of 0.5 mg Dutasteride administered once daily for 52 weeks in men with Androgenetic Alopecia types III vertex, IV and V per the Norwood-Hamilton classification. The study consists of a Screening Phase (3 weeks prior to Baseline) and a Treatment Phase (52 weeks). A subject who completes the full course of study treatment and the final study visit (Week 52; Visit 7) will be considered as study completion.

ELIGIBILITY:
Inclusion Criteria:

* Male outpatient, 20 to 50-years-old, inclusive (at the time of obtaining consent).
* AGA classified as Type III vertex, IV, or V (excluding Type IV anterior and V anterior) utilizing the Norwood-Hamilton classification.
* Fluent and literate in Japanese with the ability to comprehend and record information on the PAS SFI and DLQI questionnaires.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2 x upper limit of normal (ULN); alkaline phosphatase and bilirubin <=1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Willing to comply with study requirements, including maintaining the same hair color and hairstyle throughout the study- a) subjects who use hair colorants/hair dyes may continue to do so; however, there should be no traces of hair color remaining on the scalp at the time of study visits. b) hair length in nonbalding areas should be >=2 cm (0.75 inch) around the vertex region of the head at the time of study visits.
* Able to swallow and retain oral medication

Exclusion Criteria:

* Evidence of hypogonadism defined as serum testosterone <250 Nanogram/decilitre (ng/dl) at Screening.
* Unstable liver disease (chronic stable hepatitis B and C are acceptable if subject otherwise meets entry criteria).
* History of renal insufficiency or Serum creatinine >1.5 x ULN at Screening.
* History of malignancy within the past 5 years, except basal cell or squamous cell carcinoma of the skin.
* History of prostate cancer before the age of 50 years in a first degree relative.
* Serum PSA level >2.0 nanogram/millilitre (ng/mL) at Screening.
* History of breast cancer or clinical breast examination suggestive of malignancy.
* Active unstable thyroid disease, including subjects on therapy for either hyperthyroidism or hypothyroidism unless their dose of thyroid medication has been stable for at least 3 months.
* Any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to Screening; uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management, and subjects who are known to be acquired immunodeficiency syndrome [AIDS](including subjects with a diagnosis of human immunodeficiency virus (HIV) positive).
* History or current evidence of any serious and/or unstable pre-existing medical or psychiatric disorder, or other conditions that could, in the opinion of the investigator or GSK medical monitor, interfere with the subject's safety, obtaining informed consent, or compliance with study procedures. Note: the investigator may consult with GSK medical monitor if a condition could interfere with the subject's safety.
* Clinically relevant abnormal finding on the Screening electrocardiogram (ECG).
* Global scalp hair thinning, including occipital areas.
* Scarring of the scalp, including prior hair transplant or scalp reduction, or any other condition or disease of the scalp or hair, including diseases of the hair shaft (e.g., tinea infection, nonandrogenetic-cause of alopecia, psoriatic dermatitis or other psoriatic lesions, or uncontrolled seborrheic dermatitis).
* History of hair transplantation at any time to correct AGA or use of hair weaving within 6 months prior to Screening.
* History or evidence of hair loss other than AGA (e.g., due to an auto-immune, endocrine, mechanical or infectious process, or secondary to a scalp dermatological disorder).
* Use of any cosmetic product aimed at improving or correcting the signs of hair loss (e.g., scalp preparations with claims aiming at improved hair growth) within 2 weeks prior to Screening.
* Use of light or laser treatments on the scalp (e.g., light emitting diode [LED] lamps) within 3 months prior to Screening.
* Hypersensitivity to any 5 alpha-reductase (5AR) inhibitor or drugs chemically related to the study treatment.
* Use of Dutasteride within 18 months prior to Screening, or use of finasteride within 12 months prior to Screening.
* Previous use of systemic cytotoxic agents.
* Use of glucocorticoids (inhaled glucocorticoids are allowed; topical corticosteroids are allowed provided that they are not used on the scalp) within 3 months prior to Screening.
* Use of the following during the 6 months prior to Screening: Minoxidil (oral or topical), Carpronium chloride, Systemic drugs with anti-androgenic properties (e.g., cyproterone acetate, spironolactone, ketoconazole, flutamide, and bicalutamide). Use of ketoconazole shampoo on the scalp is prohibited during the study, but use before Screening is not a reason for exclusion. Cimetidine is prohibited during the study, but use before Screening is not a reason for exclusion, Topical estrogen or progesterone, Topical prostaglandin analogs on the scalp, Tamoxifen, Drugs potentially causing hypertrichosis (e.g., cyclosporine, diazoxide, phenytoin, psoralens), Drugs potentially causing hypotrichosis or telogen effluvium (e.g., valproic acid), Anabolic steroids, Lithium or phenothiazines.
* Participation in any investigational or marketed drug or device trial within 1 month prior to Screening for this study. Including participation in any trial for Dutasteride and administration of active drugs (Dutasteride or finasteride) prior to Screening for this study. In addition, subjects must not participate in any other drug or device trials during the course of this study.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04-14 (Actual); Primary Completion 2014-07-19 (Actual); Study Completion 2014-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tsunemi Y, Irisawa R, Yoshiie H, Brotherton B, Ito H, Tsuboi R, Kawashima M, Manyak M; ARI114264 Study Group. Long-term safety and efficacy of dutasteride in the treatment of male patients with androgenetic alopecia. J Dermatol. 2016 Sep;43(9):1051-8. doi: 10.1111/1346-8138.13310. Epub 2016 Feb 19. PMID 26893187
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114264 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male participants with androgenetic alopecia types III vertex IV and V per Norwood Hamilton classification were enrolled into study.
Pre-assignment Details: This outpatient study consisted of a Screening Phase (3 weeks prior to Baseline) and a Treatment Phase (52 weeks).
Groups:
- Dutasteride 0.5 mg: Participants received an Open-Label dutasteride 0.5 milligram (mg) capsule, Once Daily (QD) for 52 weeks.
Period: Overall Study
Arm/Group | Dutasteride 0.5 mg
Started | 120
Completed | 110
Not Completed | 10
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 120
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign(including an abnormal laboratory finding), symptom, or disease(new or exacerbated) temporally associated with the use of a medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, a congenital anomaly/birth defect, important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, drug-induced liver injury, breast cancer in male participants, prostate cancer, spontaneous abortion in female partner of male participants
Time Frame: From Baseline (Week 0) until Week 52
Population: Intent-to-Treat (ITT) Population: comprised of all participants who received a randomization number, regardless of whether or not treatment was administered
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Participants
  Any AE | 64
  Any SAE | 2

2. Primary Outcome: Number of Participants With Drug-related, Treatment-emergent AEs and AE Leading to Premature Study Drug Discontinuation and Possible Suicidality-related Adverse Event (PSRAE)
Description: An AE is considered drug-related if the relationship variable indicates so, or if the variable value is missing. Any AE with a start date on or after the treatment start date and on or before the last dose of treatment is considered on-treatment (treatment-emergent). This includes an AE with a missing onset date. Any AE which occurred, in the investigator's judgement and is possibly related to suicidality, is defined as possible suicidality-related adverse event (PSRAE). Suicidality was assessed by using the columbia-suicide severity rating scale (C-SSRS) as determined by the investigator. The C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors.
Time Frame: From Baseline (Week 0) until Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Participants
  Any drug related AEs | 20
  Any treatment-emergent AEs | 64
  Any AE leading to study drug discontinuation | 0
  Any PSRAE | 3

3. Primary Outcome: Number of Participants With Change From Baseline in Breast Examination Results Any Time Post-Baseline Visit
Description: A qualitative breast examination was performed at Baseline (Week 0), at the Week 26 Visit and at the Week 52 Visit (and at the early withdrawal visit, if applicable). Participants were assessed for presence (reported as yes) and absence (reported as no) of palpable breast tissue (PBT) or nipple tenderness (NT) and/or clinically significant (CS) PBT or NT at Baseline (BL), at each scheduled Post-BL assessment. Change from BL in breast examination results included the number of participants with change from 'no (N)' at BL to 'yes (Y)' at any Post-BL assessment for the presence of PBT or NT, and the number of participants with change from N at BL in CS to Y at any Post-BL assessment in CS for PBT and for NT. BL value of an assessment is defined as the latest assessment on or before the BL date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline to Week 52
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Participants
  PBT, Change from N at BL to Y, n=120 | 0
  PBT, CS, Y (among change from N at BL to Y), n=0 | 0
  PBT, CS, N (among change from N at BL to Y), n=0 | 0
  NT, Change from N at BL to Y, n=120 | 1
  NT, CS, Y (among change from N at BL to Y), n=1 | 1
  NT, CS, N (among change from N at BL to Y), n=0 | 0

4. Primary Outcome: Mean Change From Baseline in Hemoglobin, Albumin and Total Protein at the Indicated Time Points
Description: Blood samples were collected for the measurement of hemoglobin, albumin and total protein at Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. Change from Baseline in the hemoglobin, albumin and total protein values are summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Grams per liter (g/L)
  Hemoglobin, Week 26, n=114 | 0.61 (5.891)
  Hemoglobin, Week 52, n=111 | -0.94 (5.657)
  Hemoglobin, Final value, n=118 | -0.69 (5.792)
  Albumin, Week 26, n=114 | -0.64 (2.014)
  Albumin, Week 52, n=111 | -1.42 (1.928)
  Albumin, Final value, n=118 | -1.31 (1.969)
  Total protein, Week 26, n=114 | -0.17 (3.741)
  Total protein, Week 52, n=111 | -0.55 (3.389)
  Total protein, Final value, n=118 | -0.40 (3.415)

5. Primary Outcome: Mean Change From Baseline in Hematocrit at the Indicated Time Points
Description: Blood samples were collected for the measurement of hematocrit at Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. Change from Baseline in the hematocrit value is summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Proportion of red blood cells in blood
  Week 26, n=114 | -0.01 (0.018)
  Week 52, n=111 | 0.00 (0.019)
  Final value, n=118 | -0.00 (0.019)

6. Primary Outcome: Mean Change From Baseline in Platelet Count and White Blood Cell Count at the Indicated Time Points
Description: Blood samples were collected for the measurement of platelet count and white blood cell count at Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. Change from Baseline in the platelet count and white blood cell count values are summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter (GI/L)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
10^9 cells/Liter (GI/L)
  Platelet count, Week 26, n=114 | 3.41 (22.172)
  Platelet count,Week 52, n=109 | -1.48 (22.327)
  Platelet count,Final value, n=118 | -1.12 (22.758)
  White blood cells count, Week 26, n=114 | 0.05 (1.309)
  White blood cells count, Week 52, n=111 | 0.17 (1.269)
  White blood cells count, Final value, n=118 | 0.13 (1.197)

7. Primary Outcome: Mean Change From Baseline in Red Blood Cells Count at the Indicated Time Points
Description: Blood samples were collected for the measurement of the red blood cell count at Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. Change from Baseline in the red blood cell count value is summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
10^12 cells per liter (TI/L)
  Week 26, n=114 | -0.01 (0.200)
  Week 52, n=111 | 0.01 (0.192)
  Final value, n=118 | 0.01 (0.198)

8. Primary Outcome: Mean Change From Baseline in Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST) at the Indicated Time Points
Description: Blood samples were collected for the measurement of ALT, ALP and AST at Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. Change from Baseline in the ALT, ALP and AST values are summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Units per liter (U/L)
  ALT, Week 26, n=114 | 5.58 (13.697)
  ALT, Week 52, n=111 | 1.51 (8.516)
  ALT, Final value, n=118 | 1.14 (7.982)
  ALP, Week 26, n=114 | 0.30 (10.124)
  ALP, Week 52, n=111 | 0.24 (9.077)
  ALP, Final value, n=118 | 0.24 (9.320)
  AST, Week 26, n=113 | 4.81 (12.164)
  AST, Week 52, n=108 | 1.85 (5.263)
  AST, Final value, n=118 | 1.71 (4.982)

9. Primary Outcome: Mean Change From Baseline in Total Bilirubin and Creatinine at the Indicated Time Points
Description: Blood samples were collected for the measurement of total bilirubin and creatinine at Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. Change from Baseline in the total bilirubin and creatinine values are summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Micromoles per liter (µmol/L)
  Total bilirubin, Week 26, n=114 | -0.99 (4.495)
  Total bilirubin,, Week 52, n=111 | -0.23 (5.189)
  Total bilirubin, Final value, n=118 | -0.26 (5.302)
  Creatinine, Week 26, n=114 | -1.14 (5.525)
  Creatinine, Week 52, n=111 | 1.73 (6.514)
  Creatinine, Final value, n=118 | 1.29 (6.525)

10. Primary Outcome: Mean Change From Baseline in Potassium, Sodium, Glucose and Urea/Blood Urea Nitrogen (BUN) at the Indicated Time Points
Description: Blood samples were collected for the measurement of potassium, sodium, glucose and urea/BUN at Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. Change from Baseline in the potassium, sodium, glucose and urea/BUN values are summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Millimoles per liter (mmol/L)
  Potassium, Week 26, n=113 | 0.08 (0.289)
  Potassium,, Week 52, n=108 | 0.02 (0.308)
  Potassium, Final value, n=118 | 0.02 (0.309)
  Sodium, Week 26, n=114 | 1.22 (1.857)
  Sodium, Week 52, n=111 | 1.01 (2.143)
  Sodium, Final value, n=118 | 1.02 (2.152)
  Glucose, Week 26, n=114 | 0.48 (0.867)
  Glucose, Week 52, n=111 | 0.44 (0.822)
  Glucose, Final value, n=118 | 0.45 (0.822)
  Urea/BUN , Week 26, n=114 | 0.05 (1.175)
  Urea/BUN , Week 52, n=111 | 0.02 (1.056)
  Urea/BUN , Final value, n=118 | 0.00 (1.106)

11. Primary Outcome: Mean Change From Baseline in Prostate-specific Antigen at the Indicated Time Points
Description: Blood samples were collected for the measurement of prostate-specific antigen at Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. Change from Baseline in the prostate-specific antigen value is summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Microgram per liter (µg/L)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Microgram per liter (µg/L)
  Week 26, n=116 | -0.29 (0.550)
  Week 52, n=111 | -0.32 (0.582)
  Final value, n=118 | -0.32 (0.556)

12. Primary Outcome: Number of Participants With Any Laboratory Value Shifts From Baseline at Any Time Post-baseline
Description: Blood samples for the assessment of the indicated laboratory parameters were taken at the Baseline, Week 26 and Week 52 visits and the early withdrawal visit where applicable. The laboratory parameters included ALP, ALT, AST, total bilirubin, total protein, sodium, potassium, albumin, glucose, creatinine, urea/BUN, hemoglobin, hematocrit, red blood cell (RBC) count, platelet count, white blood cell (WBC) count, and prostate-specific antigen (PSA). A laboratory value (LV) that is within the normal range is considered normal. A LV that is above the upper limit of the normal range is considered high abnormal. A LV that is below the lower limit of the normal range is considered low abnormal. Number of participants with any LV shifts from BL at any time post-BL are presented for, normal at BL to abnormal; normal at BL to high; normal at BL to low; normal or low at BL to high; normal or high at BL to low.
Time Frame: Baseline, Week 26 and 52 visits and/or early withdrawal visit
Population: ITT Population. Only participants with a normal BL and at least one post-BL LV are analysed. ITT Population (represented by n=X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 118
Participants
  Hemoglobin, normal at BL to abnormal, n=98 | 8
  Hematocrit, normal at BL to abnormal, n=95 | 8
  Platelet count, normal at BL to abnormal, n=118 | 0
  RBC count, normal at BL to abnormal, n=99 | 11
  WBC count, normal at BL to abnormal, n=117 | 3
  Albumin, normal at BL to abnormal, n=116 | 0
  ALP, normal at BL to abnormal, n=118 | 1
  ALT, normal at BL to abnormal, n=116 | 7
  AST, normal at BL to abnormal, n=118 | 6
  Total Bilirubin, normal at BL to abnormal, n=104 | 5
  Creatinine, normal at BL to abnormal, n=99 | 10
  Glucose, normal at BL to abnormal, n=116 | 14
  Potassium, normal at BL to abnormal, n=118 | 0
  Total Protein, normal at BL to abnormal, n=118 | 2
  Sodium, normal at BL to abnormal, n=118 | 1
  Urea/BUN, normal at BL to abnormal, n=116 | 0
  PSA, normal at BL to abnormal, n=118 | 1
  Hemoglobin, normal at BL to high, n=98 | 0
  Hematocrit, normal at BL to high, n=95 | 0
  Platelet count, normal at BL to high, n=118 | 0
  RBC count, normal at BL to high, n=99 | 0
  WBC count, normal at BL to high, n=117 | 3
  Albumin, normal at BL to high, n=116 | 0
  ALP, normal at BL to high, n=118 | 1
  ALT, normal at BL to high, n=116 | 7
  AST, normal at BL to high, n=118 | 6
  Total Bilirubin, normal at BL to high, n=104 | 5
  Creatinine, normal at BL to high, n=99 | 0
  Glucose, normal at BL to high, n=116 | 14
  Potassium, normal at BL to high, n=118 | 0
  Total Protein, normal at BL to high, n=118 | 0
  Sodium, normal at BL to high, n=118 | 1
  Urea/BUN, normal at BL to high, n=116 | 0
  PSA, normal at BL to high, n=118 | 1
  Hemoglobin, normal at BL to low, n=98 | 8
  Hematocrit, normal at BL to low, n=95 | 8
  Platelet count, normal at BL to low, n=118 | 0
  RBC count, normal at BL to low, n=99 | 11
  WBC count, normal at BL to low, n=117 | 0
  Albumin, normal at BL to low, n=116 | 0
  ALP, normal at BL to low, n=118 | 0
  ALT, normal at BL to low, n=116 | 0
  AST, normal at BL to low, n=118 | 0
  Total Bilirubin, normal at BL to low, n=104 | 0
  Creatinine, normal at BL to low, n=99 | 10
  Glucose, normal at BL to low, n=116 | 0
  Potassium, normal at BL to low, n=118 | 0
  Total Protein, normal at BL to low, n=118 | 2
  Sodium, normal at BL to low, n=118 | 0
  Urea/BUN, normal at BL to low, n=116 | 0
  PSA, normal at BL to low, n=118 | 0
  Hemoglobin, normal or low at BL to high, n=118 | 0
  Hematocrit, normal or low at BL to high, n=106 | 0
  Platelet count, normal or low at BL to high, n=118 | 0
  RBC count, normal or low at BL to high, n=118 | 0
  WBC count, normal or low at BL to high, n=118 | 3
  Albumin, normal or low at BL to high, n=116 | 0
  ALP, normal or low at BL to high, n=118 | 1
  ALT, normal or low at BL to high, n=116 | 7
  AST, normal or low at BL to high, n=118 | 6
  Total Bilirubin, normal or low at BL to high n=104 | 5
  Creatinine, normal or low at BL to high, n=118 | 0
  Glucose, normal or low at BL to high, n=117 | 14
  Potassium, normal or low at BL to high, n=118 | 0
  Total Protein, normal or low at BL to high, n=118 | 0
  Sodium, normal or low at BL to high, n=118 | 1
  Urea/BUN, normal or low at BL to high, n=117 | 0
  PSA, normal or low at BL to high, n=118 | 1
  Hemoglobin, normal or high at BL to low, n=98 | 8
  Hematocrit, normal or high at BL to low, n=107 | 8
  Platelet count, normal or high at BL to low, n=118 | 0
  RBC count, normal or high at BL to low, n=99 | 11
  WBC count, normal or high at BL to low, n=117 | 0
  Albumin, normal or high at BL to low, n=118 | 0
  ALP, normal or high at BL to low, n=118 | 0
  ALT, normal or high at BL to low, n=118 | 0
  AST, normal or high at BL to low, n=118 | 0
  Total Bilirubin, normal or high at BL to low,n=118 | 0
  Creatinine, normal or high at BL to low, n=99 | 10
  Glucose, normal or high at BL to low, n=117 | 0
  Potassium, normal or high at BL to low, n=118 | 0
  Total Protein, normal or high at BL to low, n=118 | 2
  Sodium, normal or high at BL to low, n=118 | 0
  Urea/BUN, normal or high at BL to low, n=117 | 0
  PSA, normal or high at BL to low, n=118 | 0

13. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure at the Indicated Time Points
Description: Blood pressure measurements were taken to observe vital signs and included systolic blood pressure (SBP) and diastolic blood pressure (DBP) at the Screening visit, Baseline visit, Weeks 13, 26, 39, and 52 visits and the early withdrawal visit if applicable. Change from Baseline in SBP and DBP is summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline, Weeks 13, 26, 39, and 52 visits and or early withdrawal visit
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Millimeters of mercury (mmHg)
  SBP, Week 13, n=120 | -0.3 (8.80)
  SBP, Week 26, n=116 | 0.9 (9.30)
  SBP, Week 39, n=112 | 0.9 (8.70)
  SBP, Week 52, n=111 | -1.3 (9.36)
  SBP, Final value, n=120 | -1.0 (9.47)
  DBP, Week 13, n=120 | -1.3 (7.78)
  DBP, Week 26, n=116 | 1.9 (7.35)
  DBP, Week 39, n=112 | 0.4 (7.61)
  DBP, Week 52, n=111 | -0.3 (7.44)
  DBP, Final value, n=120 | -0.6 (7.50)

14. Primary Outcome: Mean Change From Baseline in Heart Rate at the Indicated Time Points
Description: Vital sign monitoring included heart rate measurement at the Screening visit, Baseline visit, Weeks 13, 26, 39, and 52 visits and the early withdrawal visit if applicable. Change from Baseline in heart rate is summarized for each post-Baseline assessment as well as for the final assessment (the last post-Baseline value in the study [final value]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date).
Time Frame: Baseline visit, Weeks 13, 26, 39, and 52 visits and or early withdrawal visit
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Beats per minute
  Week 13, n=120 | 0.3 (8.27)
  Week 26, n=116 | 0.6 (8.30)
  Week 39, n=112 | 2.7 (9.33)
  Week 52, n=111 | -0.3 (7.84)
  Final value, n=120 | -0.6 (7.87)

15. Primary Outcome: Number of Participants Experiencing Suicidal Ideation or Suicidal Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. The number of participants answering yes/no responses to questions about suicidal ideation (Question [Que] 1 and Que 2) at Baseline and post-Baseline (since last visit) and suicidal behaviors (Que 6 - Que 10) at post-Baseline (since last visit) are presented. Questions included the presence (yes) or absence (no) of the following: Que 1 - a wish to be dead; Que 2 - nonspecific (NS) active suicidal thoughts; Que 6 - preparatory acts or behavior; Que 7 - aborted attempt; Que 8 - interrupted attempt (int. att.); Que 9 - non-fatal actual suicide attempt; Que 10 - completed suicide and non-suicidal self-injurious behavior. Final assessment (FA) is the last post-Baseline measurement during the study.
Time Frame: Baseline, Week 26 and Week 52
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Participants
  BL, wish to be dead, n=103 | 2
  BL, NS active suicidal thoughts, n=103 | 0
  Week 26, wish to be dead, n=116 | 2
  Week 26, NS active suicidal thoughts, n=116 | 1
  Week 26 preparatory acts or behavior, n=116 | 0
  Week 26, aborted attempt, n=116 | 0
  Week 26, int. att., n=116 | 0
  Week 26, non-fatal actual suicide attempt, n=116 | 0
  Week 26, completed suicide, n=116 | 0
  Week 26, non-suicidal self-injurious, n=116 | 0
  Week 52, wish to be dead, n=111 | 1
  Week 52, NS active suicidal thoughts, n=111 | 0
  Week 52 preparatory acts or behavior, n=111 | 0
  Week 52, aborted attempt, n=111 | 0
  Week 52, interrupted attempt n=111 | 0
  Week 52, non-fatal actual suicide attempt, n=111 | 0
  Week 52, completed suicide, n=111 | 0
  Week 52, non-suicidal self-injurious, n=111 | 0
  FA, wish to be dead, n=118 | 3
  FA, NS active suicidal thoughts, n=118 | 1
  FA preparatory acts or behavior, n=118 | 0
  FA, aborted attempt, n=118 | 0
  FA, int. att., n=118 | 0
  FA, non-fatal actual suicide attempt, n=118 | 0
  FA, completed suicide, n=118 | 0
  FA, non-suicidal self-injurious, n=118 | 0

16. Secondary Outcome: Mean Change From Baseline (BL) in Target Area Hair Count Within a 2.54 Centimeter (cm) Diameter Circle at Week 26 and Week 52
Description: Target area hair count is based on the nonvellus hair(>= 30 micrometer[μm] in width) count within a target 2.54cm(1 inch) diameter circle at the vertex and was assessed by macrophotographic technique. A cosmetic ink dot was placed by means of a tattoo at BL on the scalp in the center of the circle as a marker to guide the placement of the hair count area at subsequent time points. If the ink dot faded between study visits, it was redone. For the macrophotography, hair was clipped before each photograph. Change from BL is defined as post-BL value minus BL value. The BL value is defined as the latest assessment on or before the BL date(latest non-missing value of either treatment start date or randomization date). The last observation carried forward(LOCF) method for missing data was used by carrying forward the last non-missing post-BL assessment value for participants with missing data and/or for participants who discontinued from the study.
Time Frame: Baseline, Week 26, and Week 52
Population: ITT Population. Only participants avilable at the specified time were analysed.
Measure: Mean (Standard Deviation); unit: Hair count
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 110
Hair count
  Week 26 LOCF | 87.3 (81.14)
  Week 52 LOCF | 68.1 (82.14)

17. Secondary Outcome: Mean Change From Baseline (BL) in Target Area Hair Width Within a 2.54 cm Diameter Circle at Week 26 and Week 52
Description: Target area hair width was based on the total width of the nonvellus hairs(>=30μm in width) within a target 2.54cm(1 inch) diameter circle at the vertex and was assessed by macrophotographic technique. A cosmetic ink dot was placed by means of a tattoo at BL on the scalp in the center of the circle as a marker to guide the placement of the hair count area at subsequent time points. If the ink dot faded between study visits, it was redone. For the macrophotography, hair was clipped before each photograph. Change from BL is defined as the post-BL value minus the BL value. The BL value of an assessment is defined as the latest assessment on or before the BL date(latest non-missing value of either the treatment start date or the randomization date). The LOCF method for missing data was used by carrying forward the last non-missing post-BL assessment value for participants with missing data and/or for participants who discontinued from the study.
Time Frame: Baseline, Week 26, and Week 52
Population: ITT Population. Only participants avilable at the specified time were analysed.
Measure: Mean (Standard Deviation); unit: microns x 10^-3
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 110
microns x 10^-3
  Week 26 LOCF | 6.7 (4.80)
  Week 52 LOCF | 6.5 (5.29)

18. Secondary Outcome: Mean Change From Baseline (BL) in Terminal Hair Count Within a 2.54 cm Diameter Circle at Week 26 and Week 52
Description: Terminal hair count was based on the terminal hair(>=60 μm in width) count within a target 2.54cm(1 inch) diameter circle at the vertex and was assessed by macrophotographic technique. A cosmetic ink dot was placed by means of a tattoo at BL on the scalp in the center of the circle as a marker to guide the placement of the hair count area at subsequent time points. If the ink dot faded between study visits, it was redone. For the macrophotography, hair was clipped before each photograph. Change from BL is defined as the post-BL value minus the BL value. BL value of an assessment is defined as the latest assessment on or before the BL date(latest non-missing value of either the treatment start date or the randomization date). The LOCF method for missing data was used by carrying forward the last non-missing post-BL assessment for participants with missing data and/or for participants who discontinued from the study.
Time Frame: Baseline, Week 26 and Week 52
Population: ITT Population. Only participants avilable at the specified time were analysed.
Measure: Mean (Standard Deviation); unit: Hair count
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 110
Hair count
  Week 26 LOCF | 60.8 (70.22)
  Week 52 LOCF | 76.9 (86.19)

19. Secondary Outcome: Mean of Median Score for Panel Global Assessment of Improvement From Baseline to 26 Weeks and 52 Weeks for Vertex and Frontal Views
Description: A central panel of 3 dermatologists independently assessed change in hair growth from Baseline to Week 26 and Week 52 using a 7-point scale: greatly decreased (-3), moderately decreased (-2), slightly decreased (-1), no change (0), slightly increased (1), moderately increased (2), and greatly increased (3). The median score, across the 3 panel members, is summarized. This assessment was performed by comparing the global photographs obtained at Baseline (Screening) with those subsequently obtained at Week 26 and Week 52. This assessment was made separately based on the global photography of the vertex and frontal views. The LOCF method for missing data was used for the assessment, if a participants was missing the Week 26 global photograph, but has a global photograph from an earlier assessment (i.e., a withdrawal visit), then that photograph was assessed during the panel review.
Time Frame: Baseline, Week 26 and Week 52
Population: ITT Population. Only participants avilable at the specified time were analysed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 117
Scores on a scale
  Week 26 LOCF, vertex view | 1.34 (0.921)
  Week 26 LOCF, frontal view | 1.21 (0.963)
  Week 52 LOCF, vertex view | 1.50 (0.897)
  Week 52 LOCF, frontal view | 1.40 (0.974)

20. Secondary Outcome: Number of Participants With the Indicated Change From Baseline (BL) in the Stage of Androgenic Alopecia (AGA) According to the Norwood-Hamilton Scale at 26 Weeks and 52 Weeks
Description: The investigator/designee assessed the stage (Stage I to Stage VII) of AGA (i.e., male pattern baldness [MPB]) by utilizing the Norwood-Hamilton scale, used to measure the progression of MPB. Stage VII indicates worse balding than Stage I. Assessment was made by direct visual examination (aided by pictures) of the participant at Screening (Baseline), Week 26, and Week 52. "v," vertex; most of the hair loss (commonly seen with advancing age) is on the vertex. "a," type a variant; major features are (1) the entire anterior hairline border recedes in unison; (2) there is no simultaneous balding of the vertex. The number of participants with stage changes from Baseline are summarized. The LOCF method for missing data was used by carrying forward the last non-missing post-Baseline assessment for participants with missing data and/or for participants who discontinued from the study.
Time Frame: Baseline, Week 26 and Week 52
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Participants
  Baseline BL Stage IIIv to W26 Stage I, n=53 | 0
  BL Stage IIIv to W26 Stage II, n=53 | 0
  BL Stage IIIv to W26 Stage IIa, n=53 | 2
  BL Stage IIIv to W26 Stage III, n=53 | 4
  BL Stage IIIv to W26 Stage IIIa, n=53 | 0
  BL Stage IIIv to W26 Stage IIIv, n=53 | 45
  BL Stage IIIv to W26 Stage IV, n=53 | 2
  BL Stage IIIv to W26 Stage IVa, n=53 | 0
  BL Stage IIIv to W26 Stage V, n=53 | 0
  BL Stage IIIv to W26 Stage Va, n=53 | 0
  BL Stage IIIv to W26 Stage VI, n=53 | 0
  BL Stage IV to W26 Stage I, n=46 | 0
  BL Stage IV to W26 Stage II, n=46 | 0
  BL Stage IV to W26 Stage IIa, n=46 | 0
  BL Stage IV to W26 Stage III, n=46 | 1
  BL Stage IV to W26 Stage IIIa, n=46 | 0
  BL Stage IV to W26 Stage IIIv, n=46 | 15
  BL Stage IV to W26 Stage IV, n=46 | 29
  BL Stage IV to W26 Stage IVa, n=46 | 0
  BL Stage IV to W26 Stage V, n=46 | 0
  BL Stage IV to W26 Stage Va, n=46 | 0
  BL Stage IV to W26 Stage VI, n=46 | 1
  BL Stage V to W26 Stage I, n=19 | 0
  BL Stage V to W26 Stage II, n=19 | 0
  BL Stage V to W26 Stage IIa, n=19 | 0
  BL Stage V to W26 Stage III, n=19 | 1
  BL Stage V to W26 Stage IIIa, n=19 | 0
  BL Stage V to W26 Stage IIIv, n=19 | 3
  BL Stage V to W26 Stage IV, n=19 | 10
  BL Stage V to W26 Stage IVa, n=19 | 0
  BL Stage V to W26 Stage V, n=19 | 5
  BL Stage V to W26 Stage Va, n=19 | 0
  BL Stage V to W26 Stage VI, n=19 | 0
  BL Stage IIIv to W52 Stage I, n=53 | 1
  BL Stage IIIv to W52 Stage II, n=53 | 2
  BL Stage IIIv to W52 Stage IIa, n=53 | 4
  BL Stage IIIv to W52 Stage III, n=53 | 14
  BL Stage IIIv to W52 Stage IIIa, n=53 | 0
  BL Stage IIIv to W52 Stage IIIv, n=53 | 28
  BL Stage IIIv to W52 Stage IV, n=53 | 4
  BL Stage IIIv to W52 Stage IVa, n=53 | 0
  BL Stage IIIv to W52 Stage V, n=53 | 0
  BL Stage IIIv to W52 Stage Va, n=53 | 0
  BL Stage IIIv to W52 Stage VI, n=53 | 0
  BL Stage IV to W52 Stage I, n=46 | 0
  BL Stage IV to W52 Stage II, n=46 | 1
  BL Stage IV to W52 Stage IIa, n=46 | 0
  BL Stage IV to W52 Stage III, n=46 | 0
  BL Stage IV to W52 Stage IIIa, n=46 | 0
  BL Stage IV to W52 Stage IIIv, n=46 | 19
  BL Stage IV to W52 Stage IV, n=46 | 26
  BL Stage IV to W52 Stage IVa, n=46 | 0
  BL Stage IV to W52 Stage V, n=46 | 0
  BL Stage IV to W52 Stage Va, n=46 | 0
  BL Stage IV to W52 Stage VI, n=46 | 0
  BL Stage V to W52 Stage I, n=19 | 0
  BL Stage V to W52 Stage II, n=19 | 0
  BL Stage V to W52 Stage IIa, n=19 | 0
  BL Stage V to W52 Stage III, n=19 | 2
  BL Stage V to W52 Stage IIIa, n=19 | 0
  BL Stage V to W52 Stage IIIv, n=19 | 4
  BL Stage V to W52 Stage IV, n=19 | 10
  BL Stage V to W52 Stage IVa, n=19 | 0
  BL Stage V to W52 Stage V, n=19 | 3
  BL Stage V to W52 Stage Va, n=19 | 0
  BL Stage V to W52 Stage VI, n=19 | 0

21. Secondary Outcome: Change From Baseline in Sexual Problems as Assessed by the Problem Assessment Scale of the Sexual Function Inventory (PAS SFI) at Week 13, Week 26, Week 39, and Week 52
Description: The Problem Assessment Scale of the Sexual Function Inventory (PAS SFI) questionnaire was used to assess participant-perceived problems in sexual function using 3 questions assessing problems with sex drive, erections and ejaculation. They are scored on a 5-point scale of 0 to 4 (0=big problem, 1= medium problem, 2=small problem, 3=very small problem, 4=no problem). Total scores range from 0-12. Change from Baseline in PAS SFI scores is defined as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date). The LOCF method for missing data was used by carrying forward the last non-missing post-Baseline assessment for participants with missing data and/or for participants who discontinued from the study.
Time Frame: Baseline, Week 13, Week 26, Week 39 and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Scores on a scale
  Week 13 LOCF | -0.6 (2.30)
  Week 26 LOCF | -0.7 (2.36)
  Week 39 LOCF | -0.3 (1.97)
  Week 52 LOCF | -0.3 (1.90)

22. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Dermatology Life Quality Index (DLQI) at Week 13, Week 26, Week 39, and Week 52
Description: The DLQI is a 10-item validated measure developed specifically to assess quality of life (QoL) in participants with dermatological conditions. It assesses six domains: symptoms and feelings, daily activities, leisure, work ⁄school, personal relationships, and treatment. The DLQI total is the sum of 10 questions, each ranging from 0 (unanswered/not relevant,not at all) to 3 (very much). The higher the score, the greater the impairment of (QoL). Change from Baseline in DLQI scores is defined as the post-Baseline value minus the Baseline value. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date). The LOCF method for missing data was used by carrying forward the last non-missing post-Baseline assessment for participants with missing data and/or for participants who discontinued from the study.
Time Frame: Baseline, Week 13, Week 26, Week 39, and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
Scores on a scale
  Week 13 LOCF | -0.15 (1.281)
  Week 26 LOCF | -0.25 (1.367)
  Week 39 LOCF | -0.27 (1.465)
  Week 52 LOCF | -0.23 (1.393)

23. Secondary Outcome: Serum Concentrations of Dihydrotestosterone (DHT) at Baseline, and After 26 Weeks and 52 Weeks
Description: Blood samples for DHT analysis was collected at Baseline, Week 26 and Week 52. DHT values at a lower limit of quantification (LLQ) were imputed using 1/2 LLQ. The Baseline value of an assessment is defined as the latest assessment on or before the Baseline date (latest non-missing value of either the treatment start date or the randomization date). The LOCF method for missing data was used by carrying forward the last non-missing post-Baseline assessment for participants with missing visit data and/or for participants who discontinued from the study.
Time Frame: Baseline, Week 26 and Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: nanomole per liter (nmol/L)
Arm/Group | Dutasteride 0.5 mg
Number analyzed (Participants) | 120
nanomole per liter (nmol/L)
  Baseline, n=120 | 1.55 (0.714)
  Week 26 LOCF, n=118 | 0.19 (0.518)
  Week 52 LOCF, n=118 | 0.17 (0.267)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) and non-serious adverse events (AE) are reported from the start of treatment until the last dose of treatment.
Description: SAEs and non-serious AEs are summarized for members of the ITT Population, comprised of all participants who received a randomization number, regardless of whether or not treatment was administered. This also includes AEs with missing onset date.
Arm/Group | Dutasteride 0.5 mg
Serious Adverse Events (participants affected / at risk) | 2/120
Other Adverse Events (participants affected / at risk) | 31/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride 0.5 mg (N=120)
Stress fracture (Injury, poisoning and procedural complications) | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride 0.5 mg (N=120)
Nasopharyngitis (Infections and infestations) | 18
Erectile dysfunction (Reproductive system and breast disorders) | 14
Libido decreased (Psychiatric disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.